CLINICAL TRIAL: NCT06594809
Title: Combination of Upper Extremity Proprioceptive Neuromuscular Facilitation and Scapular Stabilization in Nonspecific Chronic Neck Pain with Scapular Dyskinesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Fathy Khalil, Assistant Lecturer orthopedic department faculty of physical therapy Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Upper extremity PNF and SD
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Scapular Dyskinesis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: A triple-blinded randomized controlled trial will be conducted, ensuring that patients, the research assistant (who serves as the examiner for all patients), and the statistician are blinded to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group one (Placebo Comparator): Neck-focused training consisted of a) cervical stretching, b) craniocervical flexion, and c) cervical retraction exercises d) Manual therapy, for three sessions per week for four weeks (Yildiz et al., 2018).
  Interventions: Other: Traditional neck pain treatment
- Group two (Active Comparator): The patients will receive Traditional treatment of neck pain and Scapular stabilization exercises (Blackburn exercises).
  Interventions: Other: Traditional neck pain treatment + Blackburn scapular stabilization exercises
- Group three (Experimental): Patients will receive combination of traditional treatment of neck pain, SS (Blackburn exercises) and upper extremity PNF patterns.
  Interventions: Other: PNF

INTERVENTIONS:
Other: PNF — Upper extremity PNF exercise is an exercise method that dynamically stabilizes the scapula and affect scapular muscles activity (Witt et al., 2011). Upper extremity PNF patterns consisted of four diagonal patterns (D1 flexion, D2 flexion, D1 extension, and D2 extension) and six key components manual contact, body position, verbal cues pattern of movement, timing of movement and resistance. Patient will be at sitting position with involved side up, head, spine, and scapula in neutral
  Arms: Group three
Other: Traditional neck pain treatment — Cervical muscles stretch + Craniocervical retraction ex + Manual therapy
  Arms: Group one
Other: Traditional neck pain treatment + Blackburn scapular stabilization exercises — The patients will receive Traditional treatment of neck pain and Scapular stabilization exercises (Blackburn exercises). Blackburn exercises are one of the ways to treat scapular dyskinesia. Perform 2 sets of 20 repetitions of each exercise each session (3 sessions per week) for four weeks (panse et al .,2018). The exercise load will be 60% of the one-repetition maximum (1-RM) during the first week due to their first exposure to the exercises. The evaluation of one-repetition maximum (1-RM) will be every week for all exercises. From the second evaluation, more weight will be added (compare to the previous evaluation) to maintain the overload.
  Arms: Group two

SUMMARY:
To study the combination of upper extremity PNF patterns and SS exercises on improving neck pain, function, scapular position, and scapular muscles strength in patients with NSCNP and SD.

DETAILED DESCRIPTION:
Nonspecific chronic neck pain (NSCNP) affects between 10.4% and 21.3% of office and computer workers, making it one of the most prevalent disorders that physical therapists treat. It frequently has a significant impact on daily living and necessitates the utilization of several healthcare resources.

NSCNP caused by Various factors-such as female sex, older age, high job demands, low social/work support, ex-smoker status, and a history of lower back disorders. Among them, the working conditions of office workers cause postural misalignment in the neck and shoulder regions. Patients with nonspecific chronic neck pain display altered dynamic scapular stability during scapular orientation.

The scapular bone connects the neck and shoulder and plays a very important role in stabilizing the neck and shoulder complex. Helgadottir et al., 2011 reported that patients who suffer from neck pain have malfunctions, such as decreased clavicular retraction and upward rotation. The axioscapular muscles, including the trapezius, serratus anterior, rhomboid major and minor, and levator scapulae, are attached to the scapular bone and can attribute to movement of the neck and shoulder complex. Several studies demonstrated that tightness and weakness of the axioscapular muscles could induce scapular dyskinesia (SD), which refers to abnormal scapular position or movement. Rehabilitation of NSCNP is highly supported by physical therapy with evidence-based interventions. Massage and ischemic compression target the surrounding muscles. These techniques decrease tension build-up, which directly improves spasticity and hyper-tonicity. Scapular stabilization exercises proved to be very advantageous in rectification of mal alignment of the neck. The scapular stabilization (SS) helps to correct muscular imbalances and gives early insight for activating superficial cervical muscles to perform a normal range of motion (ROM) and restores clavicular retraction and normal symmetry of the cervical-scapular region.

However, (Sciascia & Kibler, 2022) reported that the identified maneuvers were often performed in an isolated manner with the body in horizontal (prone or supine) stationary positions could lead to a less than optimal rehabilitation outcome likely due to these exercises focusing on strength and encouragement of inefficient or improper motor patterns. Finally, if strength shouldn't be the focus, then it is possible scapular dysfunction is more likely rooted in issues related to motor control.

Proprioceptive neuromuscular facilitation (PNF) is a rehabilitation concept which is widely used by physiotherapists and described as a comprehensive rehabilitation concept, promoting motor learning, motor control, strength, and mobility. Upper extremity PNF patterns are often included in exercises thought to affect recruitment of the scapular muscles. These patterns improve both muscular strength and flexibility as well as utilize sensory cues such as cutaneous, visual, and auditory stimuli to improve neuromuscular control and function. Incorporation of Upper extremity PNF patterns into shoulder rehabilitation programs may also be effective in treatment of SD.

Up to the authors' knowledge, there are no empirical reports or randomized control trials that have compared a motor control focused program against a program that focuses on strength of scapular muscles. Therefore, the purpose of this study was to study the combined effect of upper extremity PNF patterns and SS exercises on pain, function, scapular position, and scapular muscles strength in patients with NSCNP and SD.

ELIGIBILITY:
Inclusion Criteria:

* 1- Have referred from orthopedic surgeon diagnosed with non specific chronic neck pain (NSCNP) that has been localized to the cervical and periscapular areas for at least three months.

  2- Aged from 18-40 years. 3- Having a score more than 10 on the Neck disability index (NDI). 4- Having SD according to Kibler's description. 5- BMI from 18.5 to 29.9 kg/m2.

Exclusion Criteria:

1. History of previous neck surgery.
2. Recent or old fractures.
3. Cognitive impairment and inability to understand the scale.
4. Systematic inflammatory disease e.g., rheumatoid arthritis and ankylosing spondylitis, neck pain with radiculopathy or neuropathy.
5. Scapular dyskinesia due to other pathology such as shoulder impingement.
6. A score of below 10 or above 40 points out of 50 on the NDI.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
scapular muscle strength | up to 4 weeks
  Hand-held dynamometer (HHD) (Model 01165, Lafayette Instrument Company, Indiana) is an easy and reliable device to assess isometric muscle strength for shoulder and scapular muscles in both clinical and research settings The patient will be instructed to maintain the midrange position during each muscle test as resistance was gradually applied via the HHD until the examiner matches the subject's effort Assess upper trapezius, middle trapezius, lower trapezius, and serratus anterior
Assessment of scapular posture | up to 4 weeks
  Assessment of scapular posture by lateral scapular slide test, It used to determine scapula involves measuring the distance from the inferior angle of the scapula to the nearest vertebral spinous process using a tape measure or goniometer in three positions: shoulder in neutral, shoulder at 45 degrees of coronal plane abduction with hands resting on hips, and the shoulder at 90 degrees abduction with the arms in full internal rotation.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol